CLINICAL TRIAL: NCT03759938
Title: OPtimal TIMing of Anticoagulation After Acute Ischaemic Stroke: a Randomised Controlled Trial
Brief Title: OPTIMAS: OPtimal TIMing of Anticoagulation After Acute Ischaemic Stroke : a Randomised Controlled Trial
Acronym: OPTIMAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/0316
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Acute; Atrial Fibrillation
Keywords: ischaemic stroke, atrial fibrilation
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Ischemic Stroke | interventions — N(4)-oleylcytosine arabinoside; Dabigatran; apixaban; edoxaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 1:1 ratio to intervention or control arms of the study. Participants and their physicians will not be blinded to study arm allocation.The exact timing of anticoagulation within the period specified for the allocated study arm is at the discretion of the treating physician, as is the choice of DOAC. Apart from the timing of DOAC initiation, the DOAC should be prescribed in accordance with usual clinical practice
Who Masked: Outcomes Assessor
Masking Description: The Event Adjudication Committee is a study group (of at least three members) responsible for the review of clinical events to ensure consistent, standardized, objective and unbiased results throughout all participating sites and minimise the likelihood of discrepant interpretations.
  This group consists of a panel of experts who have the relevant therapeutic area expertise, are experienced in clinical trials, and have been trained on the specific study protocol.
  The Event Adjudication Committee will centrally review events reported using all available clinical and imaging data and evaluate efficacy and/ or safety endpoints in a blinded and unbiased manner on a regular basis to ensure accurate, consistent and standardized assessments of important study events such as recurrent symptomatic ischaemic stroke, systemic embolism and death.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early initiation of DOAC (Experimental): Early initiation of any direct oral anticoagulant (DOAC) at a dose licensed for stroke prevention in AF, within four days (96hrs) of onset of acute ischaemic stroke
  Interventions: Drug: Direct oral anticoagulant (DOAC)
- Standard Initiation of DOAC (Active Comparator): Standard initiation of any DOAC at a dose licensed for stroke prevention in AF, no sooner than day 7 and no later than day 14 after the onset of acute ischaemic stroke (i.e. between 144hrs and 336hrs from onset).
  Interventions: Drug: Direct oral anticoagulant (DOAC)

INTERVENTIONS:
Drug: Direct oral anticoagulant (DOAC) — Any of the DOACs listed above may be used for treatment in either study arm. The DOAC will be supplied from normal hospital stock, using local hospital prescriptions.
  Other Names: dabigatran, apixaban, edoxaban, rivaroxaban

SUMMARY:
OPTIMAS is a large, prospective, partially blinded randomised controlled trial of early (within ≤4 days [96hrs]) or standard (between day 7 and day 14 after stroke onset) initiation of anticoagulation after stroke in patients with atrial fibrillation (AF), using any licensed dose of a direct oral anticoagulant (DOAC). The trial will use a non-inferiority gatekeeper approach to test for non-inferiority of early anticoagulation followed by a test for superiority, if non-inferiority is established.

DETAILED DESCRIPTION:
Current guidelines do not provide clear recommendations on the timing of OAC after acute AF-related stroke. Current United Kingdom (UK) guidelines for anticoagulation state that "delay for an arbitrary 2-week period is recommended" for "disabling" stroke and that anticoagulation can be started "no later than 14 days" for other strokes, at the prescriber's discretion.

OPTIMAS will investigate whether early initiation of DOAC treatment, within 4 days (96hrs) of onset, in patients with acute ischaemic stroke and AF is as effective as, or better than, standard initiation of DOAC treatment, no sooner than day 7 (>144hrs) and no later than day 14 (<336hrs) after onset, in preventing recurrent ischaemic stroke, systemic embolism and symptomatic intracranial haemorrhage (sICH)? Participants will be randomised 1:1 to the intervention or control. The exact timing of initiating treatment within each group is at the discretion of the treating clinician.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over
2. Clinical diagnosis of acute ischaemic stroke
3. AF, confirmed by any of:

   1. 12-lead ECG recording
   2. Inpatient ECG telemetry
   3. Other prolonged ECG monitoring technique (e.g. Holter monitor)
   4. Known diagnosis of atrial fibrillation verified by medical records (e.g. primary care records, letter from secondary care)
4. Eligibility to commence DOAC in accordance with approved prescribing recommendations confirmed by treating physician
5. Uncertainty on the part of the treating physician regarding early versus standard initiation of DOAC.

Exclusion Criteria:

1. Contraindication to anticoagulation:

   1. Coagulopathy or current or recent anticoagulation with vitamin K antagonist (VKA) leading to INR ≥1.7 at randomisation.
   2. Thrombocytopenia (platelets < 75 x 10⁹/L)
   3. Other coagulopathy or bleeding tendency (based on clinical history or laboratory parameters) judged to contraindicate anticoagulation by treating clinician
2. Contraindication to early anticoagulation

   1. Known presence of haemorrhagic transformation with parenchymal haematoma occupying >30% of the infarct volume and exerting significant mass effect (i.e. PH2) (NB: HI1, HI2 and PH1 are not considered contraindications)
   2. Presence of clinically significant intracranial haemorrhage unrelated to qualifying infarct
   3. Any other contraindication to early anticoagulation as judged by the treating clinician
3. Contraindication to use of DOAC:

   1. Known allergy or intolerance to both Factor Xa inhibitor and direct thrombin inhibitor
   2. Definite indication for VKA treatment e.g. mechanical heart valve, valvular AF, antiphospholipid syndrome
   3. Severe renal impairment with creatinine clearance (Cockcroft & Gault formula) <15 mL/min (i.e. 14 mL/min or less)
   4. Liver function tests ALT > 2x ULN
   5. Cirrhotic patients with Child Pugh score equating to grade B or C
   6. Patient is taking medication with significant interaction with DOAC, including:

      * Azole antifungals (e.g. ketoconazole, itraconazole)
      * HIV protease inhibitors (e.g. ritonavir)
      * Strong CYP3A4 inducers (e.g. rifampicin, phenytoin, carbamazepine, phenobarbital or St. John's Wort)
      * Dronedarone
4. Pregnant or breastfeeding women
5. Presence on acute brain imaging of non-stroke pathology judged likely to explain clinical presentation (e.g. mass lesion, encephalitis)
6. Inability for patient to be followed up within 90 days of trial entry
7. Patient or representative refusal to consent to study procedures, including the site informing GP and healthcare professional responsible for anticoagulation care of participants
8. Any other reason that the PI considers would make the patient unsuitable to enter OPTIMAS.

Note that current DOAC treatment is NOT an exclusion criterion, as long as the treating physician considers it appropriate to restart (or continue) according to the timings specified in the OPTIMAS trial protocol. Continuation of the DOAC would be recorded as a start time of zero hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3648 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of the combined incidence of:recurrent symptomatic ischaemic stroke,symptomatic intracranial haemorrhage and systemic embolism | At 90 days from randomisation
  OPTIMAS will investigate whether early initiation of DOAC treatment in patients with acute ischaemic stroke and atrial fibrillation is as effective as, or better than, standard initiation of DOAC treatment in preventing recurrent ischaemic stroke, systemic embolism and sICH.

SECONDARY OUTCOMES:
All-cause mortality | At 90 days from randomisation
  All cause mortality reported in both arms
Incidence of vascular death | At 90 days from randomisation
  Any incidence of vascular death reported in both arms
Incidence of recurrent ischaemic stroke | At 90 days from randomisation
  Any incidence of recurrent ischaemic stroke reported in both arms
Incidence of systemic embolism | At 90 days from randomisation
  Any incidence of incidence of systemic embolism reported in both arms
Incidence of venous thromboembolism (deep vein thrombosis [DVT], pulmonary embolism [PE], cerebral venous thrombosis [CVT]) | At 90 days from randomisation
  Any of Incidence of venous thromboembolism (deep vein thrombosis [DVT], pulmonary embolism [PE], cerebral venous thrombosis [CVT]) reported in both arms
Functional status assessed by the modified Rankin scale (mRS) in both arms | At 90 days from randomisation
  The Modified Rankin Scale measures the degree of disability and dependence following a stroke. The scale consists of 7 category descriptions, where 0 means no symptoms, 1 means no significant disability, 2 means slight disability, 3 means moderate disability, 4 means moderately severe disability, 5 means severe disability and 6 means death. The assessment is carried out by asking the participant or their carer about their activities of daily living.
Cognitive ability assessed by the Montreal Cognitive Assessment (MoCA) questionnaire in both arms | At 90 days from randomisation
  The Montreal Cognitive Assessment is a questionnaire widely used as a screening assessment for detecting cognitive impairment. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. An abbreviated version of the MoCA assessing attention, verbal learning, memory, executive functions/language and orientation can be performed over the phone. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. In a study and people with mild cognitive impairment (MCI) scored an average of 22.1.
Quality of life at 90 days assessed by EuroQol 5 Dimensions 5 level questionnaire [EQ-5D-5L] in both arms | At 90 days from randomisation
  The EQ-5D-5L includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. In instances in which the participant struggles with giving answers on their own, the participant's next-of-kin or a friend who knows the participant well will be asked to complete the EQ-5D-5L proxy version. The proxy is asked to rate how they think the participant would rate their own health-related quality of life, if the participant were able to communicate it. In case a proxy is not available, the research team member who was looking after the participant will complete it on their behalf.
Patient reported outcomes assessed by the Patient-Reported Outcomes Measurement Information System Global Health questionnaire (PROMIS-10) in both arms. | At 90 days from randomisation
  The PROMIS Global-10 short form consists of 10 items that assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. The scoring system of the PROMIS Global-10 allows each of the individual items to be examined separately to provide specific information about perceptions of physical function, pain, fatigue, emotional distress, social health and general perceptions of health where 0 means never experienced this problem or symptoms and 1 means always. The higher score for each response indicate better health.
Ongoing anticoagulation | At 90 days from randomisation
  Ongoing anticoagulation will be assessed based on patient self-reporting and follow up patient medical records if necessary in both arms
Time to first incidence of primary outcome component (recurrent ischaemic stroke, systemic embolism, or sICH) | At 90 days from randomisation
  Time to first incidence of primary outcome component (recurrent ischaemic stroke, systemic embolism, or sICH) reported in both arms
Length of hospital stay for stroke-related care | At 90 days from randomisation
  Length of hospital stay for stroke-related care in both arms
Health and social care resource use | At 90 days from randomisation
  Health and social care resources (assessed by a study specific questionnaire) in both arms
Incidence of symptomatic intracranial haemorrhage (sICH) | At 90 days from randomisation
  Incidence of symptomatic intracranial haemorrhage (sICH) classified according to site intracerebral haemorrhage (within the brain parenchyma); subdural haemorrhage; extradural haemorrhage; subarachnoid haemorrhage; and haemorrhagic transformation of a brain infarct, in both arms
Incidence of major extracranial bleeding | At 90 days from randomisation
  Incidence of major extracranial bleeding reported in both arms
Incidence of all major bleeding (intracranial and extracranial) | At 90 days from randomisation
  Incidence of all major bleeding (intracranial and extracranial) reported during the study period, in both arms
Incidence of clinically relevant non-major bleeding | At 90 days from randomisation
  Incidence of clinically relevant non-major bleeding reported in both arms

OTHER OUTCOMES:
Ongoing anticoagulation at 90 days | At 90 days from randomisation
  Ongoing anticoagulation at 90 days assessed by patient self-reporting and/ or follow up patient medical records if necessary.
Individual cognitive domain subscores | At 90 days from randomisation
  Individual cognitive domain subscores measured using the MoCA questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Werring, Prof, Study Chair — UCL
Locations (44):
- United Kingdom (44):
  - Bronglais General Hospital, Hywel Dda University Health Board, Aberystwyth
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Queen Elizabeth Hospital,University Hospitals Birmingham NHS Foundation, Birmingham
  - Royal Bournemouth Hospital, Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Bradford Royal Infirmary, Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Broomfield Hospital, Mid Essex Hospital Services NHS Trust, Broomfield
  - West Suffolk Hospital, West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Addenbrooke's Hospital NHS Trust, Cambridge
  - Glangwili General Hospita, Hywel Dda University Health Boardl, Carmarthen
  - St Peter's Hospital, Ashford and St. Peter's Hospitals NHS Foundation Trust, Chertsey
  - Royal Derby Hospital, University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Withybush General Hospital, Hywel Dda University Health Board, Haverfordwest
  - Wycombe Hospital, Buckinghamshire Healthcare NHS Trust, High Wycombe
  - Queen Elizabeth Hospital Kings Lynn NHS Trust, Kings Lynn
  - Leicester Royal Infirmary, University Hospitals of Leicester NHS Trust, Leicester
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Prince Philip Hospital, Hywel Dda University Health Board, Llanelli
  - The Royal London Hospital, Barts Health NHS Trust, London
  - Northwick Park Hospital, London North West Healthcare NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Charing Cross Hospital, Imperial College Healthcare NHS Trust, London
  - Luton and Dunstable University Hospital NHS Foundation Trust, Luton
  - The James Cook University Hospital, South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Milton Keynes University Hospital NHS Foundation Trust, Milton Keynes
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital University Hospitals Plymouth NHS Trust, Plymouth
  - Poole Hospital NHS Foundation Trust, Poole
  - Royal Preston Hospital, Lancashire Teaching Hospitals, Preston
  - Royal Berkshire NHS Foundation Trust, Reading
  - Salford Royal Hospital, Salford Royal NHS Foundation Trust, Salford
  - Salisbury District Hospital, Salisbury NHS Foundation Trust, Salisbury
  - Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Southend University Hospital NHS Foundation Trust, Southend-on-Sea
  - Kings Mill Hospital, Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield
  - Morriston Hospital, Swansea Bay University Health Board, Swansea
  - Torbay Hospital, Torbay and South Devon NHS Foundation, Torquay
  - Arrowe Park Hospital, Wirral University Teaching Hospital NHS Foundation Trust, Upton
  - Watford General Hospital, West Hertfordshire Hospitals NHS Trust, Watford
  - Royal Hampshire County Hospital, Hampshire Hospitals NHS Foundation Trust, Winchester
  - Wrexham Maelor Hospital, Betsi Cadwaladr University Health Board, Wrexham
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nash PS, Dehbi HM, Ahmed N, Arram L, Best JG, Balogun M, Bennett K, Bordea E, Caverly E, Chau M, Cohen H, Cullen M, Dore CJ, Engelter ST, Fenner R, Ford GA, Gill A, Hunter R, James M, Jayanthi A, Lip GYH, Massingham S, Murray ML, Mazurczak I, Ndoutoumou A, Norrving B, Philip J, Sims H, Sprigg N, Vanniyasingam T, Freemantle N, Wheeler DC, Werring DJ; OPTIMAS Investigators. Anticoagulation Timing in Acute Stroke With Atrial Fibrillation According to Chronic Kidney Disease: The OPTIMAS Trial. Stroke. 2025 Aug;56(8):1970-1979. doi: 10.1161/STROKEAHA.125.051457. Epub 2025 May 22. PMID 40402086
- [Derived] Ahmed N, Dehbi HM, Freemantle N, Best J, Nash PS, Ruffle JK, Doig D, Werring DJ. Optimal timing of anticoagulation after acute ischaemic stroke with atrial fibrillation (OPTIMAS): statistical analysis plan for a randomised controlled trial. Trials. 2025 Feb 19;26(1):58. doi: 10.1186/s13063-025-08761-6. PMID 39966982
- [Derived] Werring DJ, Dehbi HM, Ahmed N, Arram L, Best JG, Balogun M, Bennett K, Bordea E, Caverly E, Chau M, Cohen H, Cullen M, Dore CJ, Engelter ST, Fenner R, Ford GA, Gill A, Hunter R, James M, Jayanthi A, Lip GYH, Massingham S, Murray ML, Mazurczak I, Nash PS, Ndoutoumou A, Norrving B, Sims H, Sprigg N, Vanniyasingam T, Freemantle N; OPTIMAS investigators. Optimal timing of anticoagulation after acute ischaemic stroke with atrial fibrillation (OPTIMAS): a multicentre, blinded-endpoint, phase 4, randomised controlled trial. Lancet. 2024 Oct 23:S0140-6736(24)02197-4. doi: 10.1016/S0140-6736(24)02197-4. Online ahead of print. PMID 39491870
- [Derived] Best JG, Arram L, Ahmed N, Balogun M, Bennett K, Bordea E, Campos MG, Caverly E, Chau M, Cohen H, Dehbi HM, Dore CJ, Engelter ST, Fenner R, Freemantle N, Hunter R, James M, Lip GY, Murray ML, Norrving B, Sprigg N, Veltkamp R, Zaczyk I, Werring DJ; OPTIMAS investigators. Optimal timing of anticoagulation after acute ischemic stroke with atrial fibrillation (OPTIMAS): Protocol for a randomized controlled trial. Int J Stroke. 2022 Jun;17(5):583-589. doi: 10.1177/17474930211057722. Epub 2022 Jan 12. PMID 35018878